CLINICAL TRIAL: NCT02803840
Title: A Phase II Trial of Low-Dose Radiotherapy for the Palliation of Patients With Diffuse Large B-cell Lymphoma
Brief Title: Low-dose Radiotherapy for Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO-2011-14
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
Keywords: Large B-Cell; Diffuse
MeSH Terms: conditions — Lymphoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Other): DLBCL patients with indication for palliative radiotherapy
  Interventions: Radiation: Low-dose radiotherapy

INTERVENTIONS:
Radiation: Low-dose radiotherapy — 2 x 2 Gy on symptomatic sites only
  Other Names: LDRT

SUMMARY:
Patients with Diffuse Large B-cell Lymphoma with indication for palliative radiotherapy are treated with low-dose radiation (2 x 2 Gy) to the symptomatic sites only. The primary endpoint of the study is the response rate and Quality of Life of the patients (QoL).

DETAILED DESCRIPTION:
Response is planned at 21-day after completion of the treatment. Response assessment is based on the standard definitions of the World Health Organization using complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) as response assessment criteria. The efficacy of the treatment consisted of a reduction greater than 50% of the maximum diameter of the radiated mass (PR + CR). QoL is evaluated using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 3.0 version questionnaire. The QLQ-C30 questionnaire is self administered to the patients at baseline and at 21 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven diagnosis of DLBCL with indication for palliative radiotherapy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Response rate | Clinical response up to 21 days after treatment
  Clinical response is defined as reduction > 50% of maximum diameter of the radiated lesion

SECONDARY OUTCOMES:
Quality of life according to the EORTC QLQ-C30 questionnaire | The QLQ-C30 questionnaire is administered at baseline and at 21 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Furlan, MD, Principal Investigator — Centro di Riferimento Oncologico - Aviano
Locations (1):
- Centro di Riferimento Oncologico, Aviano, Pordenone, Italy

IPD SHARING:
Plan to Share IPD: No